CLINICAL TRIAL: NCT01119066
Title: A Phase II Trial of Transplants From HLA-Compatible Related or Unrelated Donors With CD34+ Enriched, T-cell Depleted Peripheral Blood Stem Cells Isolated by the CliniMACS System in the Treatment of Patients With Hematologic Malignancies and Other Lethal Hematologic Disorders
Brief Title: HLA-Compatible Related or Unrelated Donors With CD34+ Enriched, T-cell Depleted Peripheral Blood Stem Cells Isolated by the CliniMACS System in the Treatment of Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-050
Record Dates: First submitted 2010-05-04; First posted 2010-05-07 (Estimated); Results first posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2021-05

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Multiple Myeloma
Keywords: Leukemia; Multiple Myeloma; radiation; Thiotepa; cyclophosphamide; fludarabine; Clofarabine; CliniMACS device; GCSF; 10-050
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Multiple Myeloma; Leukemia | interventions — Whole-Body Irradiation; Thiotepa; Cyclophosphamide; Busulfan; Melphalan; fludarabine; Clofarabine

ARMS (4):
- Total Body Irradiation, Thiotepa and Cyclophosphamide (Experimental): Hyperfractionated total body irradiation to a dose of 1375-1500 cGy (depending on age, stage of disease and requirement of general anesthesia) with lung shielding) Thiotepa (5 mg/kg/day x 2 or 10 mg/kg/day x 1) Cyclophosphamide (60 mg/kg/day x 2) (or fludarabine 25mg/m2 x 5 if cyclophosphamide is contraindicated)
  Interventions: Radiation: total body irradiation; Drug: Thiotepa; Drug: Cyclophosphamide; Procedure: (CliniMACS) T-cell depleted PBSC Transplant
- Busulfan, Melphalan and Fludarabine (Experimental): Busulfan (0.8 mg/kg every 6 hours x 10 or 12 doses), (depending on disease) with dose modified according to pharmacokinetics Melphalan (70mg/m2/day x 2 ) Fludarabine (25mg/m2/ day x 5)
  Interventions: Drug: Busulfan; Drug: Melphalan; Drug: Fludarabine; Procedure: (CliniMACS) T-cell depleted PBSC Transplant
- Clofarabine, Melphalan and Thiotepa (Experimental): Clofarabine (20mg/m2/ day x 5) (or, for children <18 years of age, 30mg/m2/day x 5 if deemed suitable and with PI approval), Melphalan (70 mg/m2/day x 2) Thiotepa (5 mg/kg/day x 2 or 10mg/kg/day x1)
  Interventions: Drug: Thiotepa; Drug: Melphalan; Drug: Clofarabine; Procedure: (CliniMACS) T-cell depleted PBSC Transplant
- Melphalan, Fludarabine and Thiotepa (Experimental): Melphalan (70 mg/m2/day x 2) Fludarabine (25mg/m2/ day x 5 ) Thiotepa (5 mg/kg/day x 2 or 10mg/kg/day x1)
  Interventions: Drug: Thiotepa; Drug: Melphalan; Procedure: (CliniMACS) T-cell depleted PBSC Transplant

INTERVENTIONS:
Radiation: total body irradiation — dose of 1375-1500 cGy
  Arms: Total Body Irradiation, Thiotepa and Cyclophosphamide
Drug: Thiotepa — 5 mg/kg/day x 2 or 10 mg/kg/day x 1
  Arms: Clofarabine, Melphalan and Thiotepa; Melphalan, Fludarabine and Thiotepa; Total Body Irradiation, Thiotepa and Cyclophosphamide
Drug: Cyclophosphamide — 60 mg/ kg/day x 2 (or fludarabine 25mg/m2 x 5 if cyclophosphamide is contraindicated).
  Arms: Total Body Irradiation, Thiotepa and Cyclophosphamide
Drug: Busulfan — 0.8 mg/kg every 6 hours x 10 or 12 doses (depending on disease) with dose modified according to pharmacokinetics
  Arms: Busulfan, Melphalan and Fludarabine
Drug: Melphalan — 70mg/m2/day x 2
  Arms: Busulfan, Melphalan and Fludarabine; Clofarabine, Melphalan and Thiotepa; Melphalan, Fludarabine and Thiotepa
Drug: Fludarabine — 25mg/m2/ day x 5
  Arms: Busulfan, Melphalan and Fludarabine
Drug: Clofarabine — 20mg/m2/ day x 5 (or, for children <18 years of age, 30mg/m2/day x 5 if deemed suitable and with PI approval)
  Arms: Clofarabine, Melphalan and Thiotepa
Procedure: (CliniMACS) T-cell depleted PBSC Transplant

SUMMARY:
The purpose of this study is to find out the effects of using a system called CliniMACS to remove Tcells from blood stem cells. Removing T-cells may help stop a side effect called Graft-Versus-Host Disease (GVHD). Some studies have been done with CliniMACS, but the Food and Drug Administration (FDA) has not yet approved it.

ELIGIBILITY:
Inclusion Criteria:

* Malignant conditions or other life threatening disorders correctable by transplant for which CD34+ selected, T-cell depleted allogeneic hematopoietic stem cell transplantation is indicated such as:
* AML in 1st remission - for patients whose AML does not have 'good risk' cytogenetic features (i.e. t 8;21, t15;17, inv 16).
* Secondary AML in 1st remission
* AML in 1st relapse or > than or = to 2nd remission
* ALL/CLL in 1st remission clinical or molecular features indicating a high risk for relapse; or ALL/CLL > than or = to 2nd remission
* CML failing to respond to or not tolerating Imatinib or dasatinib in first chronic phase of disease; CML in accelerated phase second chronic phase or in CR after accelerated phase or blast crisis.
* Non-Hodgkins lymphoma with chemoresponsive disease in any of the following categories:

  1. intermediate or high grade lymphomas who have failed to achieve a first CR or have relapsed following a 1st remission who are not candidates for autologous transplants.
  2. any NHL in remission which is considered not curable with chemotherapy alone and not eligible/appropriate for autologous transplant.
* Myelodysplastic syndrome (MDS): RA//RARS/RCMD with high risk cytogenetic features or transfusion dependence as well as RAEB-1 and RAEB-2 and Acute myelogenous leukemia (AML) evolved from MDS, who are not eligible for transplantation and/or unable to enroll onto protocol IRB 08-008.
* Chronic myelomonocytic leukemia: CMML-1 and CMML-2.
* Multiple Myeloma with disease in the following categories:

  1. Patients with relapsed multiple myeloma following autologous stem cell transplantation who have achieved at least partial response following additional chemotherapy.
  2. Patients with high risk cytogenetics at diagnosis must have achieved a partial response following autologous stem cell transplantation. Patients must have complex karyotype, del17p, t4;14 and/or t14;16 by FISH and/or del13 by karyotyping.
* Other rare lethal disorders of Hematopoiesis and Lymphopoiesis for which a T-cell depleted transplant is indicated (e.g. hemophagocytic lymphohistiocytosis; refractory aplastic anemia or congenital cytopenias; non-SCID lethal genetic immunodeficiencies such as Wiskott Aldrich Syndrome, CD40 ligand deficiency, or ALPS, as well as refractory autoimmune cytopenias, PNH, metabolic storage diseases or heavily transfused congenital hemoglobinopathies).
* Accrual to each treatment arm will include up to 30 standard risk and 30 poor risk patients (60 patients/treatment arm) except for Regimen D, which will include 30 patients/treatment arm, all of which will be poor risk by virtue of risks of relapse and/or transplant related mortality.
* Standard risk patients will include eligible patients, as defined above, who are receiving transplants as treatment for MDS in RA//RARS/RCMD, AML in 1st or 2nd remission, ALL in 1st CR, NHL in 1st remission, MM in 1st remission, Very Good Partial Response, or 1st Partial Response or CML in the first chronic phase or 1st remission.
* All other patients, including those with treatment related malignancies and/or those who have AML derived from MDS, will have received extensive prior chemo/radiotherapy and, therefore, will be considered to be at poor risk of conditioning and transplant related morbidities, and potentially transplant related mortality. Patients with life threatening non-malignant genetic and acquired disorders will also, by virtue of their history of, optional transfusions and/or infection be considered poor risk. Stopping rules for non-relapse related mortality in these heavily treated patients are, therefore, slightly less stringent than patients in the poor risk transplant groups. Stopping rules for the principal endpoints of graft failure and GvHD are the same for all groups.

The following inclusion criteria are also required:

* Patient's age includes from birth on to < 70 years old.
* Patients may be of either gender or any ethnic background.
* Patients must have a Karnofsky (adult) or Lansky (pediatric) Performance Status > or = to 70%
* Patients must have adequate organ function measured by:

Cardiac: asymptomatic or if symptomatic then LVEF at rest must be > or = to 50% and must improve with exercise.

Hepatic: < 3x ULN AST and ≤ to 1.5 total serum bilirubin, unless there is congenital benign hyperbilirubinemia or if the hyperbilirubinemia is directly caused by the disease in which the patient is receiving a transplant (e.g. AML Chloroma obstructing the biliary tree). Patients with higher bilirubin levels due to causes other than active liver disease are also eligible with PI approval e.g. patients with PNH, Gilbert's disease or other hemolytic disorders.

Renal: serum creatinine < than or = to 1.2 mg/dl or if serum creatinine is outside the normal range, then CrCl > 40 ml/min (measured or calculated/estimated) Pulmonary: asymptomatic or if symptomatic, DLCO > or = to 50% of predicted (corrected for hemoglobin)

* Each patient must be willing to participate as a research subject and must sign an informed consent form.

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Active viral, bacterial or fungal infection
* Patient seropositive for HIV-I/II; HTLV -I/II
* Presence of leukemia in the CNS.

Donor Inclusion Criteria:

* Each donor must meet criteria outlined by institutional guidelines
* Donor should agree to undergo general anesthesia and bone marrow harvest collection if PBSC yield is inadequate or otherwise not transplantable for whatever reason.

Donor Exclusion Criteria

* If donors do not meet institutional guidelines, exclusion will be considered.

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2010-05-03 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard O'Reilly, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 patients received 2 separate transplants on each Arm A and C
Units Other Than Participants: Additional Transplant
Groups:
- Total Body Irradiation, Thiotepa and Cyclophosphamide: Hyperfractionated total body irradiation to a dose of 1375-1500 cGy (depending on age, stage of disease and requirement of general anesthesia) with lung shielding) Thiotepa (5 mg/kg/day x 2 or 10 mg/kg/day x 1) Cyclophosphamide (60 mg/kg/day x 2) (or fludarabine 25mg/m2 x 5 if cyclophosphamide is contraindicated)
  total body irradiation: dose of 1375-1500 cGy
  Thiotepa: 5 mg/kg/day x 2 or 10 mg/kg/day x 1
  Cyclophosphamide: 60 mg/ kg/day x 2 (or fludarabine 25mg/m2 x 5 if cyclophosphamide is contraindicated).
  (CliniMACS) T-cell depleted PBSC Transplant
- Busulfan, Melphalan and Fludarabine: Busulfan (0.8 mg/kg every 6 hours x 10 or 12 doses), (depending on disease) with dose modified according to pharmacokinetics Melphalan (70mg/m2/day x 2 ) Fludarabine (25mg/m2/ day x 5)
  Busulfan: 0.8 mg/kg every 6 hours x 10 or 12 doses (depending on disease) with dose modified according to pharmacokinetics
  Melphalan: 70mg/m2/day x 2
  Fludarabine: 25mg/m2/ day x 5
  (CliniMACS) T-cell depleted PBSC Transplant
- Clofarabine, Melphalan and Thiotepa: Clofarabine (20mg/m2/ day x 5) (or, for children <18 years of age, 30mg/m2/day x 5 if deemed suitable and with PI approval), Melphalan (70 mg/m2/day x 2) Thiotepa (5 mg/kg/day x 2 or 10mg/kg/day x1)
  Thiotepa: 5 mg/kg/day x 2 or 10 mg/kg/day x 1
  Melphalan: 70mg/m2/day x 2
  Clofarabine: 20mg/m2/ day x 5 (or, for children <18 years of age, 30mg/m2/day x 5 if deemed suitable and with PI approval)
  (CliniMACS) T-cell depleted PBSC Transplant
- Melphalan, Fludarabine and Thiotepa: Melphalan (70 mg/m2/day x 2) Fludarabine (25mg/m2/ day x 5 ) Thiotepa (5 mg/kg/day x 2 or 10mg/kg/day x1)
  Thiotepa: 5 mg/kg/day x 2 or 10 mg/kg/day x 1
  Melphalan: 70mg/m2/day x 2
  (CliniMACS) T-cell depleted PBSC Transplant
Period: Overall Study
Arm/Group | Total Body Irradiation, Thiotepa and Cyclophosphamide | Busulfan, Melphalan and Fludarabine | Clofarabine, Melphalan and Thiotepa | Melphalan, Fludarabine and Thiotepa
Started | 132; 1 Additional Transplant | 227; 0 Additional Transplant | 52; 1 Additional Transplant | 11; 0 Additional Transplant
Completed | 125; 1 Additional Transplant | 213; 0 Additional Transplant | 52; 1 Additional Transplant | 11; 0 Additional Transplant
Not Completed | 7; 0 Additional Transplant | 14; 0 Additional Transplant | 0; 0 Additional Transplant | 0; 0 Additional Transplant
Not completed — Withdrawal by Subject | 4 | 6 | 0 | 0
Not completed — Concern regarding adequacy of transplant cell dose | 2 | 1 | 0 | 0
Not completed — Relapse identified before transplant | 1 | 0 | 0 | 0
Not completed — Intercurrent medication condition rendered patient ineligible | 0 | 3 | 0 | 0
Not completed — Relapse identified before transplant | 0 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Body Irradiation, Thiotepa and Cyclophosphamide | Busulfan, Melphalan and Fludarabine | Clofarabine, Melphalan and Thiotepa | Melphalan, Fludarabine and Thiotepa | Total
Number analyzed (Participants) | 125 | 213 | 52 | 11 | 401
Age, Continuous [Median (Full Range); unit: years] | 30.3 [3.5 to 63.9] | 57.6 [2 to 73] | 28.1 [0.6 to 67.2] | 10 [0.8 to 67.2] | 48 [0.6 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 91 | 21 | 5 | 180
  Male | 62 | 122 | 31 | 6 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 10 | 6 | 4 | 38
  Not Hispanic or Latino | 64 | 145 | 30 | 5 | 244
  Unknown or Not Reported | 43 | 58 | 16 | 2 | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 9 | 13 | 5 | 2 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 17 | 1 | 2 | 33
  White | 94 | 176 | 41 | 6 | 317
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 7 | 5 | 1 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 125 | 213 | 52 | 11 | 401

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Durable Hematopoietic Engraftment for T-cell Depleted Transplants Fractionated by the CliniMACS System Administered After Each of the Four Disease Targeted Cytoreduction Regimens.
Time Frame: 3 years
Population: Please note 13 participants were not evaluated in the data set as they received a second or third HCT on protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Body Irradiation, Thiotepa and Cyclophosphamide | Busulfan, Melphalan and Fludarabine | Clofarabine, Melphalan and Thiotepa | Melphalan, Fludarabine and Thiotepa
Number analyzed (Participants) | 120 | 210 | 47 | 11
Participants
  Engrafted | 118 | 205 | 45 | 10
  Primary Graft Failure | 0 | 0 | 0 | 0
  Late graft failure | 1 | 5 | 2 | 1
  Not Evaluable Engraftment | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Acute and Chronic GVHD Following T-cell Depleted, CD34+ Progenitor Cell Enriched Transplants Fractionated by the CliniMACS System.
Description: Standard BMT-CTN and IBMTR systems clinical criteria as defined by Rowlings, et al will be used to establish and grade acute GvHD. Chronic GvHD will be diagnosed and graded according to the criteria of Sullivan (CIBMTR).
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Total Body Irradiation, Thiotepa and Cyclophosphamide | Busulfan, Melphalan and Fludarabine | Clofarabine, Melphalan and Thiotepa | Melphalan, Fludarabine and Thiotepa
Number analyzed (Participants) | 44 | 65 | 12 | 3
participants
  aGVHD II-IV | 34 | 60 | 10 | 2
  cGVHD, Limited | 2 | 4 | 1 | 0
  cGVHD, Extensive | 8 | 1 | 1 | 1

3. Primary Outcome: Incidence of Non-relapse Mortality (Transplant-related Mortality) Following Each Cytoreduction Regimen and a Transplant Fractionated by the CliniMACS System.
Time Frame: 3 years
Population: Please note 13 participants were not evaluated in the data set as they received a second or third HCT on protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Body Irradiation, Thiotepa and Cyclophosphamide | Busulfan, Melphalan and Fludarabine | Clofarabine, Melphalan and Thiotepa | Melphalan, Fludarabine and Thiotepa
Number analyzed (Participants) | 120 | 210 | 47 | 11
Participants
  Alive | 81 | 145 | 30 | 8
  Dead (not non-relapse mortality) | 23 | 24 | 3 | 0
  Dead (non-relapse mortality) | 16 | 41 | 14 | 3

4. Primary Outcome: Survival and Disease-free Survival (DFS)
Time Frame: at 6 months post transplant
Population: 2 patients received 2 separate transplants on each Arm A and C
Measure: Number; unit: percentage of participants
Arm/Group | Total Body Irradiation, Thiotepa and Cyclophosphamide | Busulfan, Melphalan and Fludarabine | Clofarabine, Melphalan and Thiotepa | Melphalan, Fludarabine and Thiotepa
Number analyzed (Participants) | 125 | 213 | 52 | 11
percentage of participants
  Survival | 93.3 | 92.4 | 87.2 | 90.9
  Disease Free Survival | 82.5 | 89.0 | 85.1 | 90.9

5. Primary Outcome: Survival and Disease-free Survival (DFS)
Time Frame: 1 year post transplant
Population: 2 patients received 2 separate transplants on each Arm A and C
Measure: Number; unit: % of pts at 1 year post transplant
Arm/Group | Total Body Irradiation, Thiotepa and Cyclophosphamide | Busulfan, Melphalan and Fludarabine | Clofarabine, Melphalan and Thiotepa | Melphalan, Fludarabine and Thiotepa
Number analyzed (Participants) | 125 | 213 | 52 | 11
% of pts at 1 year post transplant
  Survival | 80.8 | 83.8 | 85.1 | 81.8
  Disease free survival | 68.3 | 73.7 | 83.0 | 72.7

6. Primary Outcome: Survival and Disease-free Survival (DFS)
Time Frame: 2 years post transplant
Population: 2 patients received 2 separate transplants on each Arm A and C
Measure: Number; unit: % of pts at 2 years
Arm/Group | Total Body Irradiation, Thiotepa and Cyclophosphamide | Busulfan, Melphalan and Fludarabine | Clofarabine, Melphalan and Thiotepa | Melphalan, Fludarabine and Thiotepa
Number analyzed (Participants) | 125 | 213 | 52 | 11
% of pts at 2 years
  Survival | 68.7 | 72.1 | 63.8 | 71.6
  Disease Free Survival | 58.9 | 62.1 | 59.6 | 62.3

7. Secondary Outcome: Proportion of Patients Receiving Optimal CD3+ (<1x10^5/kg) Cell Doses the Proportion of Patients Receiving CD3+ T-cell Doses > 1x10^5/kg.
Time Frame: Up to 3 years
Population: 2 patients received 2 separate transplants on each Arm A and C. Please note 13 participants were not evaluated in the data set as they received a second or third HCT on protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Body Irradiation, Thiotepa and Cyclophosphamide | Busulfan, Melphalan and Fludarabine | Clofarabine, Melphalan and Thiotepa | Melphalan, Fludarabine and Thiotepa
Number analyzed (Participants) | 120 | 210 | 47 | 11
Participants
  CD3 Optimal | 120 | 210 | 47 | 11
  CD3 Suboptimal | 0 | 0 | 0 | 0

8. Secondary Outcome: Proportion of Patients Receiving Optimal CD34+ (> 5x10^6/kg) Cell Doses the Proportion Recurring Suboptimal Doses (< 2x10^6/kg) CD34+ Cells
Time Frame: 3 years
Population: Please note 13 participants were not evaluated in the data set as they received a second or third HCT on protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Body Irradiation, Thiotepa and Cyclophosphamide | Busulfan, Melphalan and Fludarabine | Clofarabine, Melphalan and Thiotepa | Melphalan, Fludarabine and Thiotepa
Number analyzed (Participants) | 120 | 210 | 47 | 11
Participants
  Optimal | 105 | 169 | 39 | 11
  Suboptimal | 0 | 1 | 0 | 0
  None | 15 | 40 | 8 | 0

9. Secondary Outcome: Correlation of Doses of CD34+ Progenitors and CD3+ T Cells With Engraftment
Time Frame: 3 years
Population: Please note 13 participants were not evaluated in the data set as they received a second or third HCT on protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Body Irradiation, Thiotepa and Cyclophosphamide | Busulfan, Melphalan and Fludarabine | Clofarabine, Melphalan and Thiotepa | Melphalan, Fludarabine and Thiotepa
Number analyzed (Participants) | 120 | 209 | 47 | 11
Participants
  Optimal (> 5x106/kg), Engrafted | 103 | 163 | 38 | 11
  Optimal (> 5x106/kg), Late Graft Failure | 1 | 5 | 1 | 0
  Optimal (> 5x106/kg), Not Evaluable | 1 | 0 | 0 | 0
  Suboptimal(< 2x106/kg), Engrafted | 0 | 1 | 0 | 0
  Suboptimal(< 2x106/kg), Late Graft Failure | 0 | 0 | 0 | 0
  Suboptimal(< 2x106/kg), Not Evaluable | 0 | 0 | 0 | 0
  Other(2-5X106/kg), Engrafted | 15 | 40 | 7 | 0
  Other(2-5X106/kg), Late Graft Failure | 0 | 0 | 1 | 0
  Other(2-5X106/kg), Not Evaluable | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Please note: participants were not censored from adverse event evaluation if they had a second or third transplant on protocol
Arm/Group | Total Body Irradiation, Thiotepa and Cyclophosphamide | Busulfan, Melphalan and Fludarabine | Clofarabine, Melphalan and Thiotepa | Melphalan, Fludarabine and Thiotepa
All-Cause Mortality (participants affected / at risk) | 42/120 | 71/210 | 18/47 | 3/11
Serious Adverse Events (participants affected / at risk) | 13/125 | 30/213 | 9/52 | 3/11
Other Adverse Events (participants affected / at risk) | 16/125 | 31/213 | 9/52 | 3/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Body Irradiation, Thiotepa and Cyclophosphamide (N=125) | Busulfan, Melphalan and Fludarabine (N=213) | Clofarabine, Melphalan and Thiotepa (N=52) | Melphalan, Fludarabine and Thiotepa (N=11)
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 3 | 0 | 0
Death NOS (General disorders) | 8 | 12 | 7 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Gen disorders & admin site conditions Other, spec (General disorders) | 0 | 1 | 0 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 3 | 0 | 1
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 0
Pericardial tamponade (Cardiac disorders) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 0
Sepsis (Infections and infestations) | 2 | 4 | 2 | 0
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Body Irradiation, Thiotepa and Cyclophosphamide (N=125) | Busulfan, Melphalan and Fludarabine (N=213) | Clofarabine, Melphalan and Thiotepa (N=52) | Melphalan, Fludarabine and Thiotepa (N=11)
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 0
Altered Mental Status (Psychiatric disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 3 | 0 | 0
CMV Viremia (Infections and infestations) | 0 | 1 | 0 | 0
Death NOS (General disorders) | 8 | 12 | 7 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Gen disorders & admin site conditions Other, spec (General disorders) | 0 | 1 | 0 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 3 | 0 | 1
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0
Mucositis Oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 0
Pericardial tamponade (Cardiac disorders) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 0
Sepsis (Infections and infestations) | 2 | 4 | 2 | 0
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Vasovagal Reaction (Nervous system disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT01119066/Prot_SAP_000.pdf